CLINICAL TRIAL: NCT00903422
Title: Study PMA112509, a Phase I/II Study of Eltrombopag in Thrombocytopenic Subjects With Advanced Myelodysplastic Syndrome (MDS) or Secondary Acute Myeloid Leukemia After MDS (sAML/MDS)
Brief Title: Eltrombopag Treatment of Thrombocytopenia in Subjects With Advanced Myelodysplastic Syndrome (MDS) or Secondary Acute Myeloid Leukemia After MDS (sAML/MDS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 112509
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Myelodysplastic Syndrome
Keywords: Advanced Myelodysplastic Syndrome; Thrombocytopenia; sAML/MDS; Eltrombopag; TPO-R agonist; de novo AML; Thrombopoietin; MDS; Thrombopoietin receptor agonist; secondary Acute Myeloid Leukemia after MDS; Platelets
MeSH Terms: conditions — Myelodysplastic Syndromes; Thrombocytopenia; Jacobs syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eltrombopag (Active Comparator): Eltrombopag
  Interventions: Drug: eltrombopag olamine
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: eltrombopag olamine — thrombopoietin receptor agonist
  Arms: Eltrombopag
Other: Placebo — Placebo tablets with no active pharmaceutical ingredient
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and tolerability of eltrombopag in the treatment of low platelet counts in adult subjects with advanced myelodysplastic syndrome (MDS), secondary acute myeloid leukemia after MDS (sAML/MDS), or de novo AML that are relapsed, refractory or ineligible to receive azacitidine, decitabine, intensive chemotherapy or autologous/allogeneic stem cell transplantation. This is a placebo-controlled study in which patients will receive study medication daily for 6 months, during which time the dose of study medication may be adjusted based upon individual platelet counts and bone marrow blast counts. All subjects will receive best standard of care (platelet transfusions, mild chemotherapy, cytokines, valproic acid, all-trans retinoic acid, ESAs or G-CSF) in addition to study medication. Subjects taking placebo may be allowed to crossover to eltrombopag treatment if a clinically and statistically significant improvement in bone marrow blast counts is seen in subjects treated with eltrombopag.

DETAILED DESCRIPTION:
A double-blind, randomized, placebo-controlled phase I/II study to evaluate the safety and tolerability of eltrombopag olamine, a thrombopoietin receptor agonist, administered for 6 months as oral tablets once daily in adult subjects with advanced MDS, sAML/MDS, or de novo AML. Study medication may be increased up to 300 mg (150 mg maximum dose for East Asian subjects), based upon individual platelet counts and bone marrow blast counts.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (18 years of age or older) with advanced MDS, sAML/MDS, or de novo AML with >=10% and <=50% blasts in bone marrow. Peripheral blood blast change over time should not be suggestive of highly proliferative disease (as judged by the investigator).
* Subjects must be dependent on regular platelet transfusions or have a platelet count taken within the 4 weeks prior to randomization that is <30 Gi/L.
* Subjects must be relapsed, refractory or ineligible to receive standard treatment options of azacitidine and decitabine and must be relapsed, refractory or ineligible to receive intensive chemotherapy or autologous/allogeneic stem cell transplantation. A subject may be considered relapsed/refractory to a standard treatment if it is discontinued due to lack of efficacy. For subjects ineligible for standard treatments, it is permissible to start one of these standard treatments while on study medication if the Investigator considers that the subject becomes eligible during the course of the study.
* Prior therapy with demethylating agents (azacitidine or decitabine), lenalidomide or IL-11(oprelvekin) must have been completed at least 4 weeks before Day 1; antithymocyte/antilymphocyte globulin, intensive chemotherapy, or autologous/allogeneic stem cell transplantation must have been completed at least 2 months before Day 1. If a subject must discontinue a course of therapy due to lack of efficacy, the washout periods listed above do not apply (and the patient may be screened and randomized immediately if other eligibility criteria are met).
* Subjects must have platelet count and platelet transfusion data available over a period of 4 weeks prior to randomization.
* Subjects with advanced MDS, sAML/MDS, or de novo AML must have stable disease indicated by a doubling time of peripheral blast counts >7 days during screening.
* During the 4 weeks prior to randomization, subjects must have a baseline bone marrow examination including the following:
* cytomorphology to confirm bone marrow blasts between 10-50%,
* cytogenetics (provide only most prevalent abnormal clone),

The results of the above tests are required prior to subject randomization.

* Supportive/palliative therapies such as cytokines (except for IL-11; oprelvekin), valproic acid, all-trans retinoic acid or mild chemotherapy are allowed if part of the local SOC, provided those therapies have been at a stable dose for 4 weeks. If the subject chooses to discontinue these therapies prior to study entry, they must be completed 4 weeks prior to enrollment into this study, unless the therapy is discontinued due to lack of efficacy. Erythropoiesis-stimulating agents (ESAs) in anemic subjects or granulocyte colony-stimulating factor (G-CSF) in subjects with severe neutropenia and recurrent infections are allowed during the study as per accepted standards. Subjects who enter the study on ESAs or G-CSF should continue at the same dose schedule until the optimal dose of study medication has been established.
* ECOG Status 0-3.
* Subject is able to understand and comply with protocol requirements and instructions.
* Subject has signed and dated informed consent.
* Prothrombin time (PT/INR) and activated partial thromboplastin time (aPTT) must be within 80 to 120% of the normal range at baseline.
* Adequate baseline organ function defined by the criteria below:
* total bilirubin (except for Gilbert's Syndrome) <= 1.5xULN
* ALT and AST <= 3xULN
* creatinine <= 2xULN
* albumin must not be below the lower limit of normal (LLN) by more than 20%.
* Subject is practicing an acceptable method of contraception (documented in chart). Female subjects (or female partners of male subjects) must either be of non-childbearing potential (hysterectomy, bilateral oophorectomy, bilateral tubal ligation or post-menopausal >1 year), or of childbearing potential and use 1 of the following highly effective methods of contraception (i.e., Pearl Index <1.0%) from 2 weeks prior to administration of study medication, throughout the study, and 28 days after completion or premature discontinuation from the study:
* Complete abstinence from intercourse;
* Intrauterine device (IUD);
* Two forms of barrier contraception (diaphragm plus spermicide, and for males condom plus spermicide);
* Male partner is sterile prior to entry into the study and is the only partner of the female;
* Systemic contraceptives (combined or progesterone only).

Exclusion Criteria:

* Subjects with a diagnosis of acute promyelocytic leukemia.
* History of treatment for cancer (other than MDS, sAML/MDS, or de novo AML) with systemic chemotherapy and/or radiotherapy within the last 2 years.
* History of treatment with romiplostim or other TPO-R agonists.
* Pre-existing cardiovascular disease (including congestive heart failure, New York Heart Association [NYHA] Grade III/IV), or arrhythmia known to increase the risk of thromboembolic events (e.g. atrial fibrillation), or subjects with a QTc >450 msec (QTc >480 msec for subjects with Bundle Branch Block).
* Bone marrow fibrosis that leads to an inability to aspirate marrow for assessment.
* Spleen size >14 cm (length as per ultrasound examination).
* Leukocytosis >=25,000/uL prior to Day 1 of study medication.
* Female subjects who are nursing or pregnant (positive serum or urine Beta-human chorionic gonadotropin [B-hCG] pregnancy test) at screening or pre-dose on Day 1.
* Current alcohol or drug abuse.
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.
* Active and uncontrolled infections.
* Subjects infected with Hepatitis B, C or Human Immunodeficiency Virus (HIV).
* Subjects with liver cirrhosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2009-05-14 (Actual); Primary Completion 2012-06-26 (Actual); Study Completion 2013-12-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability parameters including non-hematological laboratory Grade 3/Grade 4 toxicities, change in bone marrow blast counts from baseline and adverse events reporting. | Approximately 46 months

SECONDARY OUTCOMES:
Proportion of subjects with a baseline platelet count <20 Gi/L and an increase to >20 Gi/L and by at least 2x baseline; or a baseline platelet count between >=20-<30 Gi/L and an absolute platelet count increase to >=50 Gi/L at any time during treatment. | Approx. 46 months
Frequency and number of units of platelet transfusions during the treatment and follow-up periods for eltrombopag- and placebo-treated subjects. | approx 46 months
The incidence and severity of bleeding events, measured using the World Health Organization (WHO) Bleeding Scale, during the treatment and 4 week follow-up periods for eltrombopag- and placebo-treated subjects. | approx. 46 months
Overall survival (OS) of eltrombopag- and placebo-treated subjects. | approx. 46 months
Change in health-related quality of life as measured using the EQ-5D questionnaire. | approx. 46 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (59):
- United States (23):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Coral Springs, Florida
  - GSK Investigational Site, Lake Worth, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Camden, New Jersey
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, New Braunfels, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Arlington, Virginia
  - GSK Investigational Site, Fairfax, Virginia
  - GSK Investigational Site, Madison, Wisconsin
- Brazil (3):
  - GSK Investigational Site, Salvador, Estado de Bahia
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Rio de Janeiro
- Denmark (2):
  - GSK Investigational Site, Koebenhavn Oe
  - GSK Investigational Site, Odense C
- France (7):
  - GSK Investigational Site, Bayonne
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Bobigny
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Toulouse
- Germany (10):
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Göttingen, Lower Saxony
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Duisburg, North Rhine-Westphalia
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Berlin
- Hong Kong (2):
  - GSK Investigational Site, Hong Kong
  - GSK Investigational Site, Shatin, New Territories
- Italy (3):
  - GSK Investigational Site, Reggio Calabria, Calabria
  - GSK Investigational Site, Florence, Tuscany
  - GSK Investigational Site, Vicenza, Veneto
- GSK Investigational Site, San Juan, Puerto Rico
- GSK Investigational Site, Seoul, South Korea
- Taiwan (3):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
- United Kingdom (4):
  - GSK Investigational Site, Aberdeen
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, London

REFERENCES:
- [Background] Mavroudi I, Pyrovolaki K, Pavlaki K, Kozana A, Psyllaki M, Kalpadakis C, Pontikoglou C, Papadaki HA. Effect of the nonpeptide thrombopoietin receptor agonist eltrombopag on megakaryopoiesis of patients with lower risk myelodysplastic syndrome. Leuk Res. 2011 Mar;35(3):323-8. doi: 10.1016/j.leukres.2010.06.029. Epub 2010 Aug 4. PMID 20688394
- [Derived] Platzbecker U, Wong RS, Verma A, Abboud C, Araujo S, Chiou TJ, Feigert J, Yeh SP, Gotze K, Gorin NC, Greenberg P, Kambhampati S, Kim YJ, Lee JH, Lyons R, Ruggeri M, Santini V, Cheng G, Jang JH, Chen CY, Johnson B, Bennett J, Mannino F, Kamel YM, Stone N, Dougherty S, Chan G, Giagounidis A. Safety and tolerability of eltrombopag versus placebo for treatment of thrombocytopenia in patients with advanced myelodysplastic syndromes or acute myeloid leukaemia: a multicentre, randomised, placebo-controlled, double-blind, phase 1/2 trial. Lancet Haematol. 2015 Oct;2(10):e417-26. doi: 10.1016/S2352-3026(15)00149-0. Epub 2015 Oct 1. PMID 26686043
- See also: Results for study 112509 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112509?search=study&search_terms=112509#rs